CLINICAL TRIAL: NCT00937118
Title: Damage Control for Severe Duodenal and Combined Duodenal-Pancreatic Injuries: A Retrospective Review
Brief Title: Damage Control for Duodenal and Combined Duodenal-Pancreatic Injuries
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, John C. Mayberry, Professor of Surgery, Oregon Health and Science University
Other Study IDs: IRB # 5128
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-05

CONDITIONS: Injury of Duodenum; Pancreatic Injury
Keywords: laparotomy; duodenal injury; pancreatic injury; trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Injury Management: Patients with full thickness duodenal laceration undergoing laparotomy and surviving more then 72 hours at our level 1 trauma center in the years 1989-2009. Patients requiring pancreaticoduodenectomy were excluded.

SUMMARY:
The management of significant duodenal injuries and combined duodenal-pancreatic injuries continues to be challenging and controversial, and several techniques have been advocated over the years. One technique surgeons employ is the damage control/planned reoperation strategy. At the trauma center, the advent of damage control and other planned re-operation strategies has resulted in an evolution in the investigators management of duodenal lacerations and combined duodenal-pancreatic injuries. In this retrospective review, the investigators intend to quantify the investigators change in practice and to report its outcome compared to previous practice.

Using the OHSU Trauma Laparotomy Outcomes Database, the investigators will identify all patients receiving trauma laparotomy for a duodenal or duodenal/pancreatic injury for a period of 20 years, from 1989-2009. A number of data points will be retrieved from patients' medical records, including but not limited to grade of duodenal injury, mechanism of injury, Injury Severity Score, and others.

DETAILED DESCRIPTION:
The management of significant duodenal injuries and combined duodenal-pancreatic injuries continues to be challenging and controversial. Several techniques have been advocated over the years to prevent the dreaded complications of repair breakdown, fistulization, and intra-abdominal sepsis. These include duodenal diverticulization, triple tube ostomy, tube duodenostomy, and pyloric exclusion. These techniques are all designed to decompress, heal without undue intraluminal pressure or flow. Recently, surgeons have questioned whether aggressive adjunctive diversion is truly necessary, especially for less severe injuries, and many have noted complications associated with the reconstructions apart from the injury.

An alternative to routine diversion/decompression/exclusion is the damage control/planned reoperation strategies following laparotomy for severe visceral injuries that have become prevalent in the past two decades. Instead of performing a primary duodenal repair with enteral diversion or decompression in a single operation, many surgeons employ a surveillance and "touch-up" strategy over the course of 2-4 abdominal explorations. The abdominal fascia is not closed until the healing phase has commenced and the surgeon feels confident the repair will hold.

At the trauma center, the advent of damage control and other planned re-operation strategies as resulted in an evolution in our management of duodenal lacerations and combined duodenal-pancreatic injuries. The investigators perform noticeably fewer decompression, diversion, or exclusion procedures and have increasingly relied on serial abdominal explorations for surveillance of the repair.

In this retrospective review, we intend to quantify our change in practice and to report its outcome compared to previous practice.

Using the OHSU Trauma Laparotomy Outcomes Database, we will identify all patients receiving trauma laparotomy in which a duodenal or combined duodenal-pancreatic injury was identified in a 20-year period from 1989-2009. The medical records of these patients will be reviewed to confirm duodenal injury and to tabulate other factors.

The patients will be categorized based on management of the duodenal injury, e.g. primary repair, decompression, diversion, or exclusion. Patients will also be categorized according to laparotomy strategy, e.g. damage control, planned reoperation, or primary fascial closure without planned reoperation. Duodenal-related complications will be tabulated and the various groups compared. The investigators anticipate including up to 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients who received a trauma laparotomy for a duodenal or combined duodenal/pancreatic injury

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients who received a trauma laparotomy for a duodenal or combined duodenal/pancreatic injury
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Mayberry, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Stone HH, Fabian TC. Management of duodenal wounds. J Trauma. 1979 May;19(5):334-9. doi: 10.1097/00005373-197905000-00006. PMID 448769
- [Background] Snyder WH 3rd, Weigelt JA, Watkins WL, Bietz DS. The surgical management of duodenal trauma. Precepts based on a review of 247 cases. Arch Surg. 1980 Apr;115(4):422-9. doi: 10.1001/archsurg.1980.01380040050009. PMID 7362449
- [Background] Kashuk JL, Moore EE, Cogbill TH. Management of the intermediate severity duodenal injury. Surgery. 1982 Oct;92(4):758-64. PMID 7123496
- [Background] Rickard MJ, Brohi K, Bautz PC. Pancreatic and duodenal injuries: keep it simple. ANZ J Surg. 2005 Jul;75(7):581-6. doi: 10.1111/j.1445-2197.2005.03351.x. PMID 15972052
- [Background] Talving P, Nicol AJ, Navsaria PH. Civilian duodenal gunshot wounds: surgical management made simpler. World J Surg. 2006 Apr;30(4):488-94. doi: 10.1007/s00268-005-0245-0. PMID 16547621
- [Background] Seamon MJ, Pieri PG, Fisher CA, Gaughan J, Santora TA, Pathak AS, Bradley KM, Goldberg AJ. A ten-year retrospective review: does pyloric exclusion improve clinical outcome after penetrating duodenal and combined pancreaticoduodenal injuries? J Trauma. 2007 Apr;62(4):829-33. doi: 10.1097/TA.0b013e318033a790. PMID 17426536
- [Background] Rotondo MF, Schwab CW, McGonigal MD, Phillips GR 3rd, Fruchterman TM, Kauder DR, Latenser BA, Angood PA. 'Damage control': an approach for improved survival in exsanguinating penetrating abdominal injury. J Trauma. 1993 Sep;35(3):375-82; discussion 382-3. PMID 8371295
- [Background] Rotondo MF, Zonies DH. The damage control sequence and underlying logic. Surg Clin North Am. 1997 Aug;77(4):761-77. doi: 10.1016/s0039-6109(05)70582-x. PMID 9291979
- [Background] Moore EE, Burch JM, Franciose RJ, Offner PJ, Biffl WL. Staged physiologic restoration and damage control surgery. World J Surg. 1998 Dec;22(12):1184-90; discussion 1190-1. doi: 10.1007/s002689900542. PMID 9841741
- [Result] Mayberry J, Fabricant L, Anton A, Ham B, Schreiber M, Mullins R. Management of full-thickness duodenal laceration in the damage control era: evolution to primary repair without diversion or decompression. Am Surg. 2011 Jun;77(6):681-5. PMID 21679632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inpatients requiring laparotomy for trauma with duodenal injury years 1989 - 2009
Period: Overall Study
Arm/Group | Injury Management
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Injury Management
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Duodenal-related Complications
Description: Duodenal-related complications including leak, obstruction, and abscess
Time Frame: 20 years
Population: Patients with duodenal related complications
Measure: Number; unit: percentage of subjects
Groups:
- No Diversion Decompression or Exclusion: Patients with full thickness duodenal laceration undergoing laparotomy who did not have diversion, decompression, or exclusion techniques
- Diversion Decompression or Exclusion: Patients with full thickness duodenal laceration undergoing laparotomy who did have diversion, decompression, or exclusion techniques
- Damage Control: Patients with full thickness duodenal laceration undergoing laparotomy who had a damage control technique
- Fascial Closure: Patients with full thickness duodenal laceration undergoing laparotomy who did not have damage control and instead had primary fascial closure
Arm/Group | No Diversion Decompression or Exclusion | Diversion Decompression or Exclusion | Damage Control | Fascial Closure
Number analyzed (Participants) | 23 | 18 | 25 | 16
percentage of subjects | 13 | 11 | 8 | 19

ADVERSE EVENTS:
Arm/Group | Injury Management
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No